CLINICAL TRIAL: NCT05407753
Title: Effect of Oral Ketone Administration on Cognitive Function, Musculoskeletal Damage and Hormonal and Metabolic Dysregulations Induced by Ultra-endurance Running
Brief Title: Effect of Exogenous Ketosis During Ultra-endurance Exercise
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Peter Hespel, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: S65311
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Exercise; Ultra-endurance Running; Ketosis; Skeletal Muscle; Cognitive Function
MeSH Terms: conditions — Motor Activity; Ketosis | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone ester (Experimental): Subjects receive the ketone ester (R)-3-hydroxybutyl (R)-3-hydroxybutyrate (25g before ultrarun, 12.5g every 30 min during race, 25g immediately after race, 25g before sleep, 3 x 25g on day after race.
  Interventions: Dietary Supplement: Ketone ester
- Con (Placebo Comparator): Subjects receive a non-caloric, taste matched placebo (water and sucrose octaacetate).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone ester — Subjects receive the ketone ester at the following timepoints: 25g before ultrarun, 12.5g every 30 min during race, 25g immediately after race, 25g before sleep, 3 x 25g on day after race.
  Arms: Ketone ester
Dietary Supplement: Placebo — Subjects receive a non-caloric taste-matched placebo (water with sucrose octaacetate)
  Arms: Con

SUMMARY:
The aim of this study is to investigate the effect of oral ketone administration during and immediately after an ultramarathon. Potential changes in cognitive function (reaction time, number of errors), running performance, jump height, skeletal muscle inflammatory infiltration and hormonal alterations will be the main focus. In this context, subjects (n=24) will perform a 100km ultrarunning trail, while receiving either ketone ester (KE, n =12) or placebo (CON, n=12). Experimental measurements will be performed immediately before and after the ultramarathon as well as 24h after the ultramarathon.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18 and 55 years old
* Recreational or competitive runner having performed an ultramarathon (>42km) during the last 2 years
* Good health status confirmed by a medical screening
* Body Mass Index (BMI) between 18 and 25

Exclusion Criteria:

* Any kind of injury/pathology that is a contra-indication to perform ultra-endurance exercise
* Intake of any medication or nutritional supplement that is known to affect exercise performance
* Intake of analgesics, anti-inflammatory agents, or supplementary anti-oxidants, from 2 weeks prior to the start of the study.
* Blood donation within 3 months prior to the start of the study
* Smoking
* More than 3 alcoholic beverages per day
* Current participation in another research trial
* Any other argument to believe that the subject is unlikely to successfully complete the full study protocol
* Adherence to a high-fat, low-carbohydrate ketogenic diet (less than 20% of energy intake derived from carbohydrates)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-10-24 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Reaction time | Before race - immediately after race
  Change in reaction time during a reaction time task
Countermovent jump | Before race - immediately after race - 48 hours after start of race
  Change in countermovement jump height
Exercise performance | Immediately after race
  Time needed to complete the ultrarun
Skeletal muscle inflammatory cell infiltration | Before race - 48 hours after start of race
  Change in infiltration of inflammatory cells in skeletal muscle

SECONDARY OUTCOMES:
Catecholamines in blood | Before race - immediately after race - 48 hours after start of race
  Change in catecholamine concentration in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Research Group, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No